CLINICAL TRIAL: NCT01252979
Title: Ketones & Mitochondrial Heteroplasmy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Mary Kay Koenig, Principle Investigator, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-10-0091
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: MELAS Syndrome; Mitochondrial Diseases
Keywords: MELAS; Ketones; Medium Chain Triglycerides; MCT oil; Mitochondrial Disorder; Heteroplasmy; 3243AG; Subject is informed and given ample opportunity to consider his/her participation and has given his/her written consent.; Subject is willing and able to comply with all trial requirements.; Subject harbors the 3243 A>G mtDNA mutation at a level detectable in blood.; Female subjects of child-bearing potential must not be pregnant.; Subjects must not have Diabetes Mellitus.
MeSH Terms: conditions — MELAS Syndrome; Mitochondrial Diseases; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medium Chain Triglyceride (Experimental)
  Interventions: Dietary Supplement: Medium-Chain Triglycerides

INTERVENTIONS:
Dietary Supplement: Medium-Chain Triglycerides — Subjects will take supplemental MCT oil 3 times a day for 6 months

SUMMARY:
The current study is a prospective evaluation of the ability of ketosis to shift mitochondrial DNA (mtDNA) heteroplasmy in subjects harboring a known mutation in their mtDNA at position 3243 (A>G). Subjects will be given supplemental medium chain triglycerides (MCTs) for a period of 6 months. mtDNA heteroplasmy will be measured 3 months prior to treatment, at treatment initiation, and 6 months after initiation.

The primary objective of the current study is to determine if there is a shift in heteroplasmy in patients harboring the 3243 A>G mtDNA mutation to a more favorable (higher wild-type) profile while in a state of ketosis.

DETAILED DESCRIPTION:
The current study is a prospective evaluation of the ability of ketosis to shift mitochondrial DNA (mtDNA) heteroplasmy in subjects harboring a known pathogenic mutation in their mtDNA at position 3243 (A>G). Subjects will be induced in to ketosis by administration of supplemental medium chain triglycerides (MCTs) for a period of 6 months. mtDNA heteroplasmy will be assessed 3 months prior to treatment, at treatment initiation, and 6 months after initiation.

The primary objective of the current study is to determine if there is a shift in heteroplasmy in patients harboring the 3243 A>G mtDNA mutation to a more favorable (higher wild-type) genotypic profile while in a state of ketosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is informed and given ample opportunity to consider his/her participation and has given his/her written consent.
2. Subject is willing and able to comply with all trial requirements.
3. Subject harbors the 3243 A>G mtDNA mutation at a level detectable in blood.
4. Female subjects of child-bearing potential must not be pregnant. Female subjects of child-bearing potential (not surgically sterile or 2 years post-menopausal) must also agree to use appropriate contraceptive methods (abstinence, oral, injectable, implantable, or barrier) for the duration of the trial.
5. Subject must not have diabetes mellitus.

Exclusion Criteria:

1. Subject is currently participating or has participated within the last 2 months in any clinical trial involving treatment of mitochondrial disorders with MCT supplementation or induction of ketosis.
2. Subject has a medical condition that could reasonably be exacerbated by ketone supplementation (including diabetes mellitus).
3. Subject is unable to give reasonable informed consent/assent.
4. Subject is a pregnant or nursing female.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Heteroplasmy | 9 months
  Blood samples will be used to measure the degree of mitochondrial DNA heteroplasmy

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States